CLINICAL TRIAL: NCT01703689
Title: Impact of Either Audit and Feedback Only or Audit and Feedback Associated to Cooperative Work Meetings Between Hospital Geriatricians and Nursing Home Staff on Quality Indicators and Health Care Practices in Nursing Homes.
Brief Title: Impact of Educational and Professional Supportive Interventions on Nursing Home Quality Indicators
Acronym: IQUARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agence Régionale de la Santé - Midi Pyrénées (Other Government)
Collaborators: Observatoire Régional de la Santé Midi-Pyrénées (ORSMIP) (Unknown)
Responsible Party: Principal Investigator, Yves Rolland, MD PhD, University Hospital, Toulouse
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ARSMP.2010.1
Record Dates: First submitted 2012-09-27; First posted 2012-10-10 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Quality Indicators; Physical Disability
Keywords: Quality indicators; quality of care; nursing home; long-term care unit; nursing home organisation; nursing home structure; disability; dependence; functional decline; functional impairment; older adults; elderly; audit and feedback; cooperative work; geriatrician; medication; hospitalisation; comorbidity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- strong intervention group (SIG) (Experimental): Nursing homes that received audit and feedback information on quality indicators and benefited of cooperative work meetings with hospital geriatricians
  Interventions: Behavioral: Audit and Feedback; Behavioral: Cooperative Work
- intervention group (LIG) (Active Comparator): Nursing homes that only received audit and feedback information on quality indicators
  Interventions: Behavioral: Audit and Feedback

INTERVENTIONS:
Behavioral: Audit and Feedback — Descriptive statistics to each nursing home (NH) with regards to its own indicators of quality and residents' health status, and the same descriptive statistics on the sub-regional and regional levels were done to all NHs for comparative purposes.
Behavioral: Cooperative Work — Nursing homes (NH)in the strong intervention group had two half-day meetings of cooperative work with a hospital geriatrician to identify NHs' weaknesses regarding quality of care and to establish strategies for overcoming these weaknesses.
  Arms: strong intervention group (SIG)

SUMMARY:
Introduction: Efficacy of audit and feedback interventions on nursing home (NH)quality indicators is not well-established.

The main objective: The main purpose of the IQUARE study was to examine the impact of two types of audit and feedback interventions on NH quality indicators and on residents dependence levels in a 18-month follow-up.

Study hypothesis: We hypothesised that audit and feedback associated to educational and professional supportive interventions are more efficacy in improving NH quality indicators than audit and feedback only.

Secondary objectives: Investigate the impact of the interventions on

1. Residents:

   * Functional decline rate
   * Drug prescriptions (quantity and quality)
   * Prevalence of adverse health outcomes (e.g., falls)
2. NHs:

   * Planning and implementation of therapeutic measures

DETAILED DESCRIPTION:
IQUARE is a multicentric individually-tailored controlled trial comparing two types of audit and feedback interventions:

* audit and feedback associated to cooperative work meetings between hospital geriatricians and nursing home (NH) staff in a 6-month intervention (strong intervention)
* audit and feedback only (light intervention) Power statistics and sample size calculations indicated that each group should be composed of at least 2 500 individuals. The strong intervention will last 6 months and is composed of two face-to-face cooperative meetings (hospital geriatricians and NH staff). Data will be collected at baseline and in a 18-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes (NH) voluntarily accepted to participate in the study.
* NH residents of both sex
* Residents living in the NH for ≥ 30 days
* Residents and their general practitioner (GP) having received information about the study
* NH residents do not voluntarily decline to participate in the study

Exclusion Criteria:

* NH currently participating in another interventional study
* GP of NH residents refused participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8039 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in nursing home quality indicators at 18 months | baseline and 18-month follow-up
  Indicators of quality of care in 10 main outcomes: dementia (e.g.,prevalence of cognitive assessment), behavioural disturbances (e.g., prevalence of behavioural disturbances assessment), restraining (e.g., prevalence of restrained residents with a medical prescription for restraining), mood (e.g., prevalence of mood assessment), osteoporosis and falls (e.g., systematic analysis of fall records), nutrition (e.g., prevalence of residents who were weighed ≥ 3 times in the last 3 months), pressure ulcers (e.g., prevalence of residents who were evaluated for the risk of pressure ulcers), pain (e.g., prevalence of residents who were evaluated for pain among residents in end-of-life), medication (e.g., prevalence of re-evaluation of residents' drug prescriptions among residents who take psychotropic), and care and services (e.g., prevalence of hospitalisations in the emergency department in the last 12 months).

SECONDARY OUTCOMES:
Onset of dependence in activities of daily living from baseline to 18 months follow-up | baseline and 18-month follow-up
  Onset of dependence will be measured using the 6-item Katz ADL scale. Activities examined are: bathing, dressing, transferring, walking inside home, incontinence, and eating/drinking. Ability in executing each activity will be set as: "able to execute alone, without difficulty", "able to execute alone, with some difficulty", or "needing help to execute or unable to execute".

OTHER OUTCOMES:
Reduction in the prescription of psychotropic drugs from baseline to 18-month follow-up | baseline and 18-month follow-up
  It will be examined if the rate of antidepressants, anxiolytics, antipsychotics, and hypnotics/sedatives (coded according to the Anatomical Therapeutic Chemical classification. Information available at: http://www.whocc.no/atc_ddd_index/) prescriptions will be reduced between baseline and follow-up. A particular attention will be given to the prevalence of people taking 3 or more psychotropics (increased risk of drug-drug interaction and adverse drug reaction) and to the use of these medications among people with dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Rolland, MD, PhD, Principal Investigator — La Grave- Casselardit University Hospital Centre, Service de Médecine Interne et Gérontologie Clinique - Gérontopôle
Locations (175):
- France (175):
  - EHPAD le parc ALBI, Albi
  - EHPAD Canarie Vieuzac, Argelès-Gazost
  - MAPAD Les Pradels, Assier
  - Les Jardins auscitains, Auch
  - Les jardins d´Agape, Auch
  - Saint Dominique, Auch
  - EHPAD Résidence Mutualiste La Pyrénéenne, Aureilhan
  - EHPAD Résidence Castelmouly, Bagnères-de-Bigorre
  - ONAC résidence paul oddo, Barbazan
  - Korian Les Ainés du Lauragais, Baziege
  - Notre Dame, Beaumont-de-Lomagne
  - Ehpad Sherpa, Belmont-sur-Rance
  - Le Pastel, Bessières
  - Le Pastourel, Bessières
  - Sainte-Cécile, Bessières
  - Emeraude, Blagnac
  - Résidence de Vinci, Blagnac
  - EHPAD St joseph de BRASSAC, Brassac
  - EHPAD Robert Durrieu, Bretenoux
  - M.R Orpea, Cahors
  - EHPAD La Cascade, Cajarc
  - Les Roses, Calmont
  - EHPAD Gai Logis, Capdenac-Gare
  - EHPAD La Croix Bleue, Capdenac-Gare
  - EHPAD le bosc Carmaux, Carmaux
  - Tour Tottier, Castelginest
  - La Cerisaie, Castelmaurou
  - Notre Dame du Bon Accueil, Castelnau-d´Estrétefonds
  - M.R St Luc - Castelnau Montratier, Castelnau-Montratier
  - Chic Ehpad C.H, Castelsarrasin
  - EHPAD Villégiale Saint Jacques CHIC - CASTRES/MAZAMET, Castres
  - MAPA Résidence St Astier, Catus
  - EHPAD Caylus - Val de Bonnette, Caylus
  - EHPAD Arc-En-Ciel, Cazals
  - Jeanne Penent, Cazères
  - Castelgirou, Cépet
  - ALLIANCE, Cologne
  - EHPAD St Laurent, Cruéjouls
  - EHPAD les arcades, Dourgne
  - EHPAD Saint-Philippe, Ercé
  - Saint-Joseph, Fronton
  - EHPAD St ANDRE CH de Gaillac, Gaillac
  - EHPAD St JEAN CH de Gaillac, Gaillac
  - EHPAD Accueil du Frère Jean, Galan
  - EHPAD La Baïse, Galan
  - Ch Gimont, Gimont
  - Foyer Pierre Bonhomme, Gramat
  - MR Charles de Gaulle, Gramat
  - MR Louis Conte, Gramat
  - EHPAD Saint Dominique, Gramond
  - Ehpad de Graulhet, Graulhet
  - Saint-Jacques, Grenade
  - Ste Sophie, Grisolles
  - EHPAD Résidence Zélia, Ibos
  - EHPAD Le Jonquère, Juillan
  - EHPAD Faux-Bourg Saint-Adrien, L'Isle-en-Dodon
  - Saint-Jacques, L'Isle-Jourdain
  - EHPAD Gustave Pédoya, La Bastide-de-Sérou
  - EHPADRouanet-Iché de LABASTIDE-ROUAIROUX, Labastide-Rouairoux
  - EHPADL'Oustal d'En Thibaud, Labruguière
  - M.R La Miséricorde, Lacapelle-Marival
  - EHPAD St vinçent de paul, Lacaune
  - Résidence du Lac, Lafrançaise
  - EHPAD résidence le grand champ, Lagrave
  - Les Causeries, Laguépie
  - Centre hospitalier du Pays d´Olmes - Laroques d´Olmes, Laroques d´Olmes
  - La Barbacane, Larrazet
  - MAPAD Les Ségalines, Latronquière
  - Résidence Paul et Lisa, Launaguet
  - Ehpad Les Quietudes, Lautrec
  - Centre hospitalier du Pays d´Olmes - Résidence du Touyre, Lavelanet
  - La Vendinelle, Le Cabanial
  - Ehpad Barrere, Lectoure
  - Ehpad Feral, Lectoure
  - Résidence Curtis, Léguevin
  - EHPAD L´Oasis, Livinhac-le-Haut
  - EHPAD La Madone, Lourdes
  - EHPAD Le Petit Jer, Lourdes
  - EHPAD Notre Dame des Grâces, Lugan
  - EHPAD Le Paginet, Lunac
  - MAPAD Les logis de l´Impernal, Luzech
  - EHPAD Le santoulis, Luzenac
  - EHPAD Saint Joseph, Marcillac-Vallon
  - Val de Gers, Masseube
  - EHPAD Le Clos du Raunier, Mazères
  - MR Beau Séjour, Mercuès
  - EHPAD du CH Millau - St Michel, Millau
  - EHPAD Les Charmettes, Millau
  - EHPAD Louise de Roquelaure, Mirepoix
  - EHPAD de MONESTIES, Monestiés
  - Ange Gardien, Montauban
  - Montauban - Ehpad Ushpa, Montauban
  - MR Saint Orens, Montauban
  - St Jean Marie Vianney, Montbeton
  - MR Sainte-Marie, Montcuq
  - M.R La Roseraie, Montfaucon
  - MR L´Etoile du Soir, Montredon
  - L´Hermitage, Montréjeau
  - EHPAD Rés. Parc de la Corette, Mur-de-Barrez
  - Le Barry, Muret
  - Résidence Marie-Antoinette, Muret
  - EHPAD Résidence les deux vallées, Nant
  - EHPAD Sainte Marie les Ursulines, Nant
  - EHPAD Résidence du Lac, Orleix
  - Centre Alzheimer Marie-Louise, Pechbonnieu
  - La Houlette, Pibrac
  - La Tranquilité, Pins-Justaret
  - Cité Saint Joseph, Plaisance Du Gers
  - Le Prat, Plaisance-du-Touch
  - Oasis-Palmeraie, Pointis-de-Rivière
  - EHPAD La résidence du Lac, Pont-de-Salars
  - L´Auta, Portet-sur-Garonne
  - EHPAD Résidence du petit bois, Pradines
  - M.R Les balcons du Lot, Prayssac
  - M.R Les Lavandes, Puy-l´Évêque
  - EHPAD la Maison Du Lac, Puygouzon
  - Résidence Isatis, Quint-Fonsegrives
  - EHPAD Hermitage et Terrasses de Rabastens, Rabastens
  - EHPAD de Revel, Revel
  - EHPAD Jean Baptiste Delfau, Réquista
  - EHPAD Les Rosiers, Rignac
  - Bel Adour, Riscle
  - EHPAD Bon Accueil, Rodez
  - EHPAD Julie Chauchard, Rodez
  - EHPAD Saint Cyrice, Rodez
  - EHPAD Saint Jacques du CH, Rodez
  - EHPAD Le clos de Siloe, Roquecourbe
  - EHPAD La Miséricorde, Saint-Affrique
  - Les Clos des Amandiers, Saint-Alban
  - EHPAD St Jean, Saint-Amans-des-Cots
  - Résidence de l´abbaye, Saint-Antonin-Noble-Val
  - Lavallée, Saint-Clar
  - EHPAD Les Galets d´Olt, Saint-Côme-d´Olt
  - Le Mas Saint-Pierre, Saint-Gaudens
  - L´Ensoleillade, Saint-Gaudens
  - EHPAD de l´Hôpital local, Saint-Geniez-d'Olt
  - Centre hospitalier Ariège Couserans, Saint-Girons
  - EHPAD Le Val d´Olt, Saint-Laurent-d'Olt
  - EHPAD Hector d´Ossun, Saint-Lizier
  - Les Rossignols, Saint-Lys
  - Maréchal Leclerc, Saint-Lys
  - Résidence La Joie de Vivre, Saint-Lys
  - EHPAD Clos St François, Saint-Sernin-sur-Rance
  - Ehpad Chez Nous, Saint-Sulpice
  - EHPAD Les grands chênes, Saïx
  - EHPAD Petite Plaisance SAVAGNAC, Salvagnac
  - EHPAD Vert Coteau, Saverdun
  - EHPAD Paul Ané, Seix
  - La Septfontoise, Septfonds
  - Ehpad Le Pre Fleuri, Serviès
  - EHPAD Sainte Marie, Siradan
  - EHPAD St Vinçent et Ste Croix, Sorèze
  - Les Tourelles, Toulouse
  - Maurice Garrigou, Toulouse
  - Plénitude Saint-Michel, Toulouse
  - Résidence Saint-Simon, Toulouse
  - La Cotonnière, Toulouse
  - Arc-en-Ciel, Toulouse
  - EHPAD Les Fontaines, Toulouse
  - La Pastellière, Toulouse
  - Orpéa Crampel, Toulouse
  - Caroline Baron, Toulouse
  - Le Grand Marquisat, Tournefeuille
  - Ehpad Belcantou, Trébas
  - EHPAD Résidence Les Rives du Pélam, Trie-sur-Baïse
  - EHPAD du Centre Hospitalier Des Deux Rives, Valence
  - M.R Résidence Valpré, Vayrac
  - EHPAD ND de Touscayrats, Verdalle
  - MR Saint Jacques, Verdun-sur-Garonne
  - EHPAD La Clairière - Les Acacias, Vic-en-Bigorre
  - Ch Vic-Fezensac, Vic-Fezensac
  - Le Château fleuri, Vic-Fezensac
  - EHPAD Sainte Claire, Villefranche-de-Rouergue
  - EHPAD Sud Rulhedu CH, Villefranche-de-Rouergue
  - Le Pin, Villeneuve-Tolosane

REFERENCES:
- [Derived] Dubucs X, de Souto Barreto P, Rolland Y. Organizational and environmental factors associated with transfers of nursing home residents to emergency departments. Eur Geriatr Med. 2018 Jun;9(3):339-346. doi: 10.1007/s41999-018-0059-x. Epub 2018 May 8. PMID 34654246
- [Derived] Cool C, Cestac P, McCambridge C, Rouch L, de Souto Barreto P, Rolland Y, Lapeyre-Mestre M. Reducing potentially inappropriate drug prescribing in nursing home residents: effectiveness of a geriatric intervention. Br J Clin Pharmacol. 2018 Jul;84(7):1598-1610. doi: 10.1111/bcp.13598. Epub 2018 May 14. PMID 29607568
- [Derived] Laffon de Mazieres C, Lapeyre-Mestre M, Vellas B, de Souto Barreto P, Rolland Y. Organizational Factors Associated With Inappropriate Neuroleptic Drug Prescribing in Nursing Homes: A Multilevel Approach. J Am Med Dir Assoc. 2015 Jul 1;16(7):590-7. doi: 10.1016/j.jamda.2015.01.092. Epub 2015 Mar 10. PMID 25769961